CLINICAL TRIAL: NCT07231783
Title: A Confirmatory, Randomised, Double-Blind, Placebo-Controlled, Parallel Study to Assess the Effects of a Dietary Supplement Containing Urolithin A (Mitopure®) on Muscle Strength and Performance in Healthy Middle-Aged Adults
Brief Title: The Effect of Urolithin A (Mitopure®) Supplementation on Muscle Strength in Healthy Middle-Aged Adults
Acronym: ATLAS 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AFCRO-197
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Healthy Aging; Muscle Function
Keywords: Urolithin A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- 500 mg Mitopure® (Experimental)
  Interventions: Dietary Supplement: Mitopure® 500mg
- 1000 mg Mitopure® (Experimental)
  Interventions: Dietary Supplement: Mitopure® 1000mg

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo softgels
  Arms: Placebo
Dietary Supplement: Mitopure® 500mg — Softgels providing 500 mg of Mitopure®
  Arms: 500 mg Mitopure®
Dietary Supplement: Mitopure® 1000mg — Softgels providing 1000 mg of Mitopure®
  Arms: 1000 mg Mitopure®

SUMMARY:
This is a randomised, double-blind, placebo-controlled, parallel study to assess the effects of Urolithin A (Mitopure®) supplementation on muscle strength and performance in healthy middle-aged adults. Participants will be randomized to consume Mitopure® (500 mg), Mitopure® (1000 mg), or placebo once daily for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Be able to give written informed consent.
* 2. Be between 40 to 65 years of age, inclusive.
* 3. Has a BMI between 25.0 and 34.9 kg/m2.
* 4. Low physical activity levels as assessed by the International Physical Activity Questionnaire (IPAQ).
* 5. Participants with low VO2 peak (defined as <35 mL/kg/min via the ergometer prior to baseline).
* 6. Willing to avoid exercising 48-h prior to study visits and maintain low physical activity status for the duration of the study.
* 7. Willing to avoid caffeine and other stimulants (e.g., energy drinks) 12-h before exercise as per study guidelines.
* 8. Willing to consume the Study Product daily for the duration of the study.

Exclusion Criteria:

* 1. Participants who are pregnant or wish to become pregnant during the study or who are lactating and/or currently breastfeeding.
* 2. Participants currently of biological childbearing potential, but not using a continuous effective method of contraception, as outlined below:

  * a. Complete abstinence from intercourse two weeks prior to administration of the Study Product, throughout the clinical study, until the completion of follow-up procedures or for two weeks following discontinuation of the Study Product in cases where Participant discontinues the study prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding two weeks when they present to the clinic for the final visit).
  * b. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that Participant.
  * c. Sexual partner(s) is/are exclusively female.
  * d. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm), tubal ligation, or contraceptive pill. The Participant must be using this method for at least one week prior to and one week following the end of the study.
  * e. Use of any intrauterine device (IUD) or contraceptive implant. The Participant must have the device inserted at least two weeks prior to the first screening visit, throughout the study, and two weeks following the end of the study.
* 3. Participants with history of drug and/or alcohol abuse at the time of enrolment. (Drinks more than nationally recommended units per week (>11 units for women; >17 units for men); alcohol/substance abuse disorder).
* 4. Participants consuming large quantities of pomegranate juice or walnuts or frequent consumers of raspberries, strawberries or cloudberries (2-week washout).
* 5. Chronic nicotine use.
* 6. Participants who are unable to swallow capsules.
* 7. Is hypersensitive to or has dietary restrictions for any of the components of the Study Product e.g., gelatine
* 8. Unstable body weight or recent participation in a weight loss program (within 12-weeks prior to screening).
* 9. Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results. Excluded health conditions include:

  * a. Major illness/surgery in the 12-weeks prior to screening
  * b. Diagnosed cardiovascular disease (NHYA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmia, uncontrolled hypertension)
  * c. Diagnosed liver disease (cirrhosis, end stage liver disease)
  * d. Diagnosed kidney disease (stage 3b or 4 chronic kidney disease, or kidney failure)
  * e. Diagnosed gastrointestinal disease (IBS/IBD, diarrhoea, Acid Reflux)
  * f. Uncontrolled thyroid conditions
  * g. Uncontrolled diabetes
  * h. Metallic implants
  * i. Conditions requiring chemotherapy or immunotherapy.
* 10. Current or recent use of a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited medications include:

  * a. Statins or other medications known to impair mitochondrial function.
  * b. Anxiolytics, antidepressants, sedative hypnotics (in the 8 weeks prior to visit 1)
  * c. Antipsychotics, monoamine Oxidase Inhibitors (in the 8 weeks prior to visit 1)
  * d. Oral anti- infective (antibiotics, antivirals, antifungals) for acute infections (in the 12-weeks prior to visit 1)
  * e. Proton pump inhibitors (PPIs) (in the 4 weeks prior to visit 1)
  * f. Corticosteroids (> 5mg per day in the past 4 weeks prior to visit 1)
  * g. GLP-1 agonists (in the 8 weeks prior to visit 1)
* 11. Current or recent (in the past 6-weeks prior to Visit 1) use of prohibited nutritional or non-nutritional supplements that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited supplements include:

  * a. Mitopure® containing supplements
  * b. Supplements for muscle strengthening/building or mitochondrial boosting supplements (e.g. high protein, Vitamin B3 [and precursors], L-carnitine, CoQ10, NAD+, resveratrol)
* 12. Blood donation in the 8-weeks prior to screening.
* 13. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
* 14. Participants may not be participating in other clinical studies. If the participant has previously taken part in an experimental study (physical or muscle performance), the Investigator must ensure sufficient time has elapsed before entry to this study to ensure the integrity of the results.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum isokinetic knee flexion strength | 6 months
  Change in maximum isokinetic knee flexion strength between Mitopure® groups and placebo measured by Biodex dynamometry (unit: Nm)

SECONDARY OUTCOMES:
Maximum isokinetic knee flexion strength | 4 months
  Change in maximum isokinetic knee flexion strength between Mitopure® groups and placebo measured by Biodex dynamometry (unit: Nm)
Maximum isokinetic knee extension strength | 4, 6 months
  Change in maximum isokinetic knee extension strength between Mitopure® groups and placebo measured by Biodex dynamometry (unit: Nm)
Maximum isometric knee flexion strength | 4, 6 months
  Change in maximum isometric knee flexion strength between Mitopure® groups and placebo measured by Biodex dynamometry (unit: Nm)
Maximum isometric knee extension strength | 4, 6 months
  Change in maximum isometric knee extension strength between Mitopure® groups and placebo measured by Biodex dynamometry (unit: Nm)
Maximum shoulder flexion strength | 4, 6 months
  Change in maximum shoulder flexion strength between Mitopure® groups and placebo measured by Biodex dynamometry (unit: Nm)
Maximum shoulder extension strength | 4, 6 months
  Change in maximum shoulder extension strength between Mitopure® groups and placebo measured by Biodex dynamometry (unit: Nm)
Body composition (lean mass) | 4, 6 months
  Change in lean mass between Mitopure® groups and placebo measured by dual-energy X-ray absorptiometry (unit: kg)
Physical performance (vertical jump) | 4, 6 months
  Change in physical performance between Mitopure® groups and placebo measured by maximum vertical jump height (unit: cm)

OTHER OUTCOMES:
Cardiovascular fitness (VO2max) | 4, 6 months
  Change in cardiovascular fitness (VO2max) between Mitopure® groups and placebo measured by a graded exercise test (unit: mL/kg/min)
Physical capacity (time to exhaustion) | 4, 6 months
  Change in physical capacity between Mitopure® groups and placebo measured by time to exhaustion during the graded exercise test (unit: minutes)
Physical capacity (maximum cycling distance) | 4, 6 months
  Change in physical capacity between Mitopure® groups and placebo measured by maximum cycling distance during the graded exercise test (unit: meters)
Physical performance (30-second chair stand) | 4, 6 months
  Change in physical performance between Mitopure® groups and placebo measured by the 30-second chair stand test (unit: repetitions)
Physical performance (6-minute walk test) | 4, 6 months
  Change in physical performance between Mitopure® groups and placebo measured by the 6-minute walk test (unit: meters)
Physical performance (timed up-and-go) | 4, 6 months
  Change in physical performance between Mitopure® groups and placebo measured by the timed up-and-go test (unit: seconds)
Blood acylcarnitine level | 6 months
  Change in blood acylcarnitine level between Mitopure® groups and placebo
Blood inflammation level | 6 months
  Change in blood inflammatory markers (TNF-alpha, IL-6, hsCRP) between Mitopure® groups and placebo
Plasma Urolithin A level | 6 months
  Change in plasma Urolithin A level between Mitopure® groups and placebo
Habitual dietary intake | 4, 6 months
  Change in habitual dietary intake between Mitopure® groups and placebo measured by 3-day diet diary
Habitual physical activity | 4, 6 months
  Change in habitual physical activity between Mitopure® groups and placebo measured by the International Physical Activity Questionnaire
Daily fatigue | 4, 6 months
  Change in self-reported daily fatigue between Mitopure® groups and placebo measured by FACIT-Fatigue questionnaire
Safety (adverse events) | 6 months
  Adverse events monitored throughout trial

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No